CLINICAL TRIAL: NCT00634946
Title: A Multicenter, Randomized, Double-blind Recommended Dose-finding Study of SI-6603 in Patients With Lumbar Disc Herniation (Phase II/III Study)
Brief Title: SI-6603 Versus Placebo in Patients With Lumbar Disc Herniation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seikagaku Corporation (Industry)
Responsible Party: Takao Murayama, Clinical Development Dept., Research & Development Div.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6603/1021; 6603/1021
Record Dates: First submitted 2008-02-27; First posted 2008-03-13 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Lumbar Vertebra Hernia
Keywords: Chemonucleolysis; Lumbar Vertebrae; Hernia
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- I (Experimental)
  Interventions: Drug: SI-6603
- II (Experimental)
  Interventions: Drug: SI-6603
- III (Experimental)
  Interventions: Drug: SI-6603
- IV (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SI-6603 — SI-6603 is administrated into the nucleus pulposus of an intervertebral disc.
  Arms: I; II; III
Drug: Placebo — Placebo is administrated into the nucleus pulposus of an intervertebral disc.
  Arms: IV

SUMMARY:
The purpose of this study is to determine whether SI-6603 is effective in the treatment of lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lumbar disc herniation (L4-L5 or L5-S1) as assessed by MRI and clinical symptoms corresponding to position of the impaired nerve root
* Patients assessed as positive in the SLR test
* Patients with sciatica in either lower leg
* Patients with no improvement from pharmacotherapy or concomitant treatment with drug and nerve block

Exclusion Criteria:

* Patients who have 2 or more lumbar disc herniations as assessed by MRI
* Patients with "extrusion-type" or "sequestration-type" herniation in whom a rupture into the posterior longitudinal ligament is identified by MRI
* Patients who have received nerve block within 3 weeks before screening
* Patients who have undergone lumbar operation, chemonucleolysis, or percutaneous nucleotomy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Changes in leg pain from baseline. | 13 weeks

SECONDARY OUTCOMES:
The leg pain | At each assessment time point

CONTACTS AND LOCATIONS:
Locations (8):
- Japan (8):
  - Chugoku Area, Chugoku
  - Chubu Area, Chūbu
  - Hokkaido Area, Hokkaido
  - Kansai Area, Kansai
  - Kanto Area, Kanto
  - Kyushu Area, Kyushu
  - Shikoku Area, Shikoku
  - Tohoku Area, Tōhoku

REFERENCES:
- [Derived] Matsuyama Y, Chiba K, Iwata H, Seo T, Toyama Y. A multicenter, randomized, double-blind, dose-finding study of condoliase in patients with lumbar disc herniation. J Neurosurg Spine. 2018 May;28(5):499-511. doi: 10.3171/2017.7.SPINE161327. Epub 2018 Feb 9. PMID 29424676